CLINICAL TRIAL: NCT05342311
Title: Preoperative Ultrasonographic Evaluation of the Right Common Femoral Vein Diameter for Predicting Spinal Anesthesia-induced Hypotension in Elderly Patients. A Prospective Observational Study.
Brief Title: Preoperative Ultrasonographic Evaluation of the Right Common Femoral Vein Diameter for Predicting Spinal Anesthesia-induced Hypotension in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud AbdelKader, principal investigator, Cairo University
Other Study IDs: MD-10-2022
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Spinal Anesthesia-induced Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: preoperative ultrasonographic evaluation of right common femoral vein diameter — preoperative ultrasonographic evaluation of right common femoral vein diameter to predict spinal anesthesia-induced hypotension in elderly patients

SUMMARY:
In this study we will determine the ability of preoperative ultrasonographic evaluation of the right common femoral vein diameter to predict spinal anesthesia-induced hypotension in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or more.
* ASA score I & II.
* Patients scheduled for surgeries under spinal anesthesia.

Exclusion Criteria:

* Negative consent.
* pre-existing hypertension
* Diabetes mellitus or autonomic neuropathy.
* Emergency operations.
* Absolute contraindications or failure to perform spinal anesthesia.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: A total of 68 consecutive elderly patients, aged >65 years scheduled for elective surgical operations under spinal anesthesia will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
The sensitivity of the transverse diameter (mm) value of the right common femoral vein as measured by ultrasound before anesthesia to predict spinal aneshesia-induced hypotension in elderly patients. | 30 minutes after spinal anesthesia

SECONDARY OUTCOMES:
Incidence of spinal anesthesia-induced hypotension in elderly | 30 minutes after spinal anesthesia
The sensitivity of the peak velocity of blood flow (mm/s) in the right common femoral vein as measured by ultrasound before anesthesia to predict spinal anesthesia-induced hypotension in elderly patients | 30 minutes after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospital, Cairo, Giza Governorate, Egypt